CLINICAL TRIAL: NCT04104919
Title: A Phase 2 Randomized Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Single Intrathecal Preoperative Administration of Brivoligide Injection in Patients With a Pain Catastrophizing Scale Score ≥16 Undergoing Mastectomy With Immediate Tissue Expander or Implant Placement
Brief Title: Study to Evaluate a Preop Dose of Brivoligide Injection for Pain After Mastectomy in Patients With High PCS Scores
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Initiation delayed due to COVID 19
Sponsor: Adynxx, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADYX-006; 1UG3DA048375-01 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative
Keywords: Mastectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brivoligide Injection 660 mg/6 mL (Experimental): Subjects randomized to the brivoligide treatment group will receive a single 660 mg/6 mL intrathecal administration of brivoligide injection while in the lateral decubitus position at lumbar interspace L3/4 or higher. After injection subjects will be placed supine in a 15-degree head down tilt (Trendelenburg position) for 5 minutes and then returned to supine horizontal for surgery.
  Interventions: Drug: Brivoligide Injection 660 mg/6 mL
- Placebo 6 mL (Placebo Comparator): Subjects randomized to the placebo group will receive a single 6 mL intrathecal administration of placebo while in the lateral decubitus position at lumbar interspace L3/4 or higher. After injection subjects will be placed supine in a 15-degree head down tilt (Trendelenburg position) for 5 minutes and then returned to supine horizontal for surgery.
  Interventions: Drug: Placebo 6 mL

INTERVENTIONS:
Drug: Brivoligide Injection 660 mg/6 mL — Single preoperative intrathecal injection
  Other Names: AYX1 Injection 660 mg/6 mL
  Arms: Brivoligide Injection 660 mg/6 mL
Drug: Placebo 6 mL — Single preoperative intrathecal injection
  Arms: Placebo 6 mL

SUMMARY:
This is a multiple center, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of brivoligide injection administered intrathecally before surgery in patients with high Pain Catastrophizing Scale (PCS) scores undergoing mastectomy with immediate tissue expander or implant placement.

DETAILED DESCRIPTION:
Potential subjects will be prescreened for PCS score; pre-qualified patients will be invited to the investigative site for informed consent and full screening within 30 days of randomization. Patients providing informed consent and meeting all study eligibility criteria will be enrolled in the study on the day of surgery (Day 1).

Subjects will receive study drug just prior to anesthesia induction. Study assessments will be entered by subjects in the electronic diary from Day 1 through Day 21. Follow-up visits will occur on Days 7 and 21 (± 2 days).

ELIGIBILITY:
Inclusion Criteria:

* Score of 16 or greater on the PCS scale
* Scheduled to undergo unilateral or bilateral mastectomy with immediate tissue expander or implant placement
* American Society of Anesthesiologists Physical Status Classification System ≤ 3
* Medically stable for this surgery with general anesthesia and intrathecal administration of study drug as determined by the Investigator
* Body mass index of 18-45 kg/m2
* Have a stable medical regimen (for prescribed medications) for ≥ 7 days before randomization
* Able to read and understand study instructions in English or Spanish, and willing and able to comply with all study procedures

Exclusion Criteria:

* Prior breast surgery in the index breast (either breast for bilateral surgery) in the last two years, other than biopsies and small/moderate volume lumpectomies
* Induction chemotherapy or plans for adjunctive chemotherapy or any radiotherapy within 21 days of surgery
* Known spinal deformities or cutaneous infection in the lumbar area that would preclude intrathecal administration of study drug
* Planned use of liposomal formulated or long-acting local anesthetics, extended release opioid formulations (e.g., Oxycontin), long half-life opioids (e.g., methadone), or drugs with potential for adverse cognitive or memory effects (e.g., ketamine, scopolamine, or propranolol) preoperatively and/or at any time through the duration of the study
* Use of more than 40 mg per day (on average) of oral morphine or its equivalent within 1 month prior to randomization
* Current neurologic disorder, which could confound the assessment of pain
* Unstable mental condition which would prevent the patient from understanding the nature and scope of the study and/or evidence of an uncooperative attitude in the opinion of the Investigator
* Women who are pregnant or nursing
* Participation in a clinical trial with the last dose or intervention within 1 month of randomization, or planned treatment in a clinical trial during this study
* Previous participation in any study involving brivoligide injection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Pain with general movement involving the chest and upper body | Day 3 to Day 14
  Least Squares (LS) Mean pain rating with general movement involving the chest and upper body on the 0 - 10 Numerical Rating Scale (0 = No Pain; 10 = Worst Pain)

SECONDARY OUTCOMES:
Pain at rest | Day 3 to Day 14
  Least Squares (LS) Mean pain rating at rest on the 0 - 10 Numerical Rating Scale (0 = No Pain; 10 = Worst Pain)
Pain with deep full inspiration and forceful effective cough | Day 3 to Day 14
  Least Squares (LS) Mean pain rating with deep full inspiration and forceful effective cough on the 0 - 10 Numerical Rating Scale (0 = No Pain; 10 = Worst Pain)
Pain with ipsilateral arm abduction | Day 14 to Day 21
  Least Squares (LS) Mean pain rating with ipsilateral arm abduction on the 0 - 10 Numerical Rating Scale (0 = No Pain; 10 = Worst Pain)
Total use of postoperative opioid medications | Day 3 to Day 14
  Total use (median) of postoperative opioid medications (morphine equivalents)
Total use of postoperative opioid medications | Day 1 through Day 21
  Total use (median) of postoperative opioid medications (morphine equivalents)
Change from baseline for the BREAST-Q | Screening to Day 21
  Change from baseline to Day 21 for the BREAST-Q

IPD SHARING:
Plan to Share IPD: No